CLINICAL TRIAL: NCT01426633
Title: Phase I Dose Escalating Trial Evaluating the Combination of Gemcitabine and Trabectedin in Patients With Advanced and/or Metastatic Leiomyosarcoma or Liposarcoma
Brief Title: Combination Therapy of Gemcitabine and Trabectedin in L-sarcomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Bernd Kasper, PD Dr. med., Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GISG-02
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2014-12-16 (Estimated); Status verified 2014-12

CONDITIONS: Leiomyosarcoma; Liposarcoma
Keywords: L-sarcomas
MeSH Terms: conditions — Leiomyosarcoma; Liposarcoma | interventions — Gemcitabine; Trabectedin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Trabectedin (Experimental)
  Interventions: Drug: Gemcitabine + Trabectedin

INTERVENTIONS:
Drug: Gemcitabine + Trabectedin — Combination therapy of gemcitabine and trabectedin

SUMMARY:
L-sarcomas represent about one third of all adult soft tissue sarcomas (24 % liposarcomas and 12 % leiomyosarcomas). Approval for the induction of trabectedin into the treatment armamentarium of advanced and/or metastatic soft tissue sarcomas after treatment failure with anthracyclines and/or ifosfamide depended mainly on its activity in the L-sarcomas (Garcia-Carbonero 2004, Le Cesne 2005, and Demetri 2009). Significant activity has been described for the use of gemcitabine and especially the combination of gemcitabine and docetaxel mainly in leiomyosarcomas and liposarcomas (Maki 2007). However, the combination of gemcitabine and docetaxel is associated with significant toxicity. Pulmonary toxicity and refractory peripheral oedema are the most common severe adverse events. The aim of the present phase I study will be to examine safety data of this promising treatment combination of gemcitabine and trabectedin in L-sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed L-sarcomas (leiomyosarcoma and liposarcoma)
* Measurable disease according to RECIST 1.1
* Any treatment line except adjuvant setting: evidence of primary metastatic situation or disease progression within the last 6 months (based on RECIST 1.1) in computed tomography or magnetic resonance imaging
* Any prior treatment possible
* Age >= 18 years
* WHO PS =< 1
* Effective contraception during study medication and up to 3 months from treatment discontinuation
* Signed informed consent form

Exclusion Criteria:

* Surgical intervention < 4 weeks
* Pregnancy or lactation
* Known allergic reaction to trabectedin or gemcitabine or one of their components
* The following laboratory values:

Absolute neutrophil count < 1.5 x 103/mm3 Platelets < 100.000/mm3 Hb < 9 g/dL Serum creatinine >= 2.5 mg/dl SGOT and/or SGPT and/or alkaline phosphatase and/or CPK > 2.5 x ULN Total bilirubin > 1 x ULN except in the case of Gilbert's syndrome

* Participation in another study (four weeks before and during the study)
* Prior malignancy apart from completely resected basal cell carcinoma of the skin or carcinoma in situ of the uterine cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To assess the maximum tolerated dose (MTD) of the combination of gemcitabine and trabectedin (Yondelis®) in patients with advanced and/or metastatic leiomyosarcoma and liposarcoma. | 12 months

SECONDARY OUTCOMES:
To assess the recommended phase II dose (RPTD) of the combination of gemcitabine and trabectedin (Yondelis®) in patients with advanced and/or metastatic leiomyosarcoma and liposarcoma. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Kasper, MD, PhD, Principal Investigator — University of Heidelberg, Mannheim University Medical Center
Locations (1):
- Mannheim University Medical Center, Mannheim, Germany

REFERENCES:
- [Derived] Kasper B, Reichardt P, Pink D, Sommer M, Mathew M, Rauch G, Hohenberger P. Combination of trabectedin and gemcitabine for advanced soft tissue sarcomas: results of a phase I dose escalating trial of the German Interdisciplinary Sarcoma Group (GISG). Mar Drugs. 2015 Jan 13;13(1):379-88. doi: 10.3390/md13010379. PMID 25591040